CLINICAL TRIAL: NCT02627586
Title: High Intensity Interval Training & Early Adverse Remodelling After Left Ventricular mYocardial Infarction (HIIT-EARLY): A Randomized Controlled Exercise Intervention Study
Brief Title: High-Intensity Interval Training Early After Left Ventricular Myocardial Infarction
Acronym: HIIT-EARLY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIIT-EARLY
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Myocardial Infarction
Keywords: exercise therapy; left ventricular remodeling; ventricular ejection fraction; high-intensity interval training
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling | interventions — High-Intensity Interval Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moderate intensity continuous exercise (Active Comparator): Moderate intensity continuous exercise (MICE) is performed on a cycle ergometer at an intensity of 50-80% of peak VO2 or 60-85% of peak heart rate for 38 min (including a 5 min warm-up and 3 min cool-down). This group will perform MICE training three times per week. Cycling resistance will be adjusted weekly according to heart rate and Borg scale.
  Interventions: Other: MICE
- High-intensity interval training (Experimental): High-intensity interval training (HIIT) is performed on a cycle ergometer. It consists of a 10 min warm-up followed by 4 min intervals in Zone III (at 90-95% of peak heart rate), with each interval separated by 3 min of active pauses in zone I (at 50-70% of peak heart rate). The total duration of the HIIT training is 38 min. Moderate intensity continuous exercise (MICE) is also performed on a cycle ergometer at an intensity of 50-80% of peak VO2 or 60-85% of peak heart rate for 38 min (including a 5 min warm-up and 3 min cool-down). This group performs two HIIT sessions and one MICE session per week.
  In both training forms cycling resistance will be adjusted weekly according to heart rate and Borg scale.
  Interventions: Other: HIIT

INTERVENTIONS:
Other: HIIT — High-intensity interval training (HIIT) is performed on a cycle ergometer. It consists of a 10 min warm-up followed by 4 min intervals in Zone III (at 90-95% of peak heart rate), with each interval separated by 3 min of active pauses in zone I (at 50-60% of peak heart rate). The total duration of the HIIT training is 38 min.
  Other Names: High intensity interval training
  Arms: High-intensity interval training
Other: MICE — MICE is also performed on a cycle ergometer at an intensity of 50-80% of peak VO2 or 60-75% of peak heart rate for 47 min (in order for the two training protocols to be isocaloric). The control group will perform MICE training three times per week.
  Other Names: Moderate intensity continuous exercise
  Arms: Moderate intensity continuous exercise

SUMMARY:
Several studies have shown that high-intensity interval training (HIIT) is more effective than moderate-intensity continuous exercise training (MICE) at improving functional capacity and quality of life in stable cardiac patients and can be performed safely.

However, its effect on patients after recent myocardial infarction is currently unknown. In these patients avoidance of a negative remodeling after an acute myocardial infarction is of upmost importance. Therefore, assessment of the influence of HIIT on post-infarct left ventricular-remodeling is urgently needed.

Therefore, the aim of this study is to determine the effect of HIIT on left ventricular (LV) remodeling (measured by LV end diastolic volume) compared to the effect of the more established MICE training modality.

Further measurements include other parameters of LV remodeling (LV contractility, and brain natriuretic peptide), prognostic parameters (peak oxygen uptake, exercise capacity), cardiac output, endothelial function, leg muscle function and scores of quality of life. Further, certain blood parameters and heart rate variability measured by electro-cardiogram are measured to assess the safety of this type of training.

Patients with first ST-segment elevation myocardial infarction (STEMI) or equivalent with onset of symptoms of ischemia and treated by primary percutaneous intervention within the preceding 4 weeks will be included.

The HIIT and MICE is integrated in a 12-week exercise training program at the Inselspital Bern, consisting of 1) exercise training, 2) nutrition counselling and 3) psychotherapy. The exercise program will comprise 3 weekly exercise sessions lasting 90 minutes, supervised by experienced exercise therapists. The program focuses on endurance type exercises, strengthening and relaxation exercises as well as exercises to improve coordination skills. In the first 3 weeks (run-in-phase), all patients will complete three weekly MICE sessions. In the following 9 weeks, patients randomized to the intervention group will perform two weekly HIIT sessions and one MICE session per week. The control group will continue with three weekly MICE sessions for the 9 week intervention phase.

A total of 144 patients will be recruited. Measurements will be performed at baseline, after a 3-week run-in-phase, and after the 9-week intervention phase. Safety measurements will be performed during the 4th and 12th week.

DETAILED DESCRIPTION:
Background

Several studies have shown that high-intensity interval training (HIIT) is more effective than moderate-intensity continuous exercise training (MICE) at improving functional capacity and quality of life in stable cardiac patients and can be performed safely.

It has therefore emerged as a new and important exercise modality in cardiac rehabilitation centres all over Europe for stable heart failure patients with LV dysfunction. Its safety and efficacy has not yet been tested in patients with acute LV dysfunction due to a myocardial infarction. In clinical practice, the difference between acute and chronic left ventricular dysfunction is often not made and patients with a condition after a recent myocardial infarction and LV dysfunction might be offered the same training regimens as patients with chronic heart failure, including HIIT, although its effect on post-infarction remodeling is unknown. On the other hand, avoidance of a negative remodeling after an acute myocardial infarction is of upmost importance. Therefore, assessment of the influence of HIIT on post-infarct LV-remodeling is urgently needed.

Objective

To determine the effect of HIIT on left ventricular remodelling (measured by end diastolic volume) compared to the effect of the more established MICE training modality in patients after a recent myocardial infarction and LV dysfunction.

Methods

After a 3-week run-in phase with MICE only training for all patients, patients randomised to the HIIT group will perform two HIIT and one MICE session per week while the MICE group performs 3 MICE sessions per week. Outcomes will be assessed before and after the 9-week intervention. End diastolic volume will be measured by 2-dimensional echography, peak oxygen uptake (peak VO2) and exercise capacity by cardiopulmonary exercise testing on a cycle ergometer, quality of life by questionnaires, vascular function by arterial stiffness measurement, leg muscle cross-sectional area by peripheral quantitative computed tomography, and leg muscle function by jumping mechanography. During the 4th and the 12th week of the rehabilitation training, heart rate variability will be measured in the morning following training, and blood samples will be taken after a training session to analyse markers of myocardial stress (Troponin T, MR-proANP, BNP).

ELIGIBILITY:
Inclusion Criteria:

* first ST-segment elevation myocardial infarction (STEMI)
* Percutaneous intervention within the preceding 4 week

Exclusion Criteria

* inability to participate in a 3-month training program
* contraindication to maximal exercise test (CPET)
* known chronic heart failure with LV ejection fraction ≤45% before the acute index event
* angiographically documented significant coronary stenosis (> 50%) at randomization
* medical condition which would prevent a patient from performing high intensity training
* permanent atrial fibrillation
* alcohol or drug abuse
* inability to follow the procedures of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-11-11 (Actual)

PRIMARY OUTCOMES:
Left ventricular end diastolic volume | week 12
  Standard transthoracic echocardiography will be performed. Left ventricular (LV) volumes will be calculated using the biplane Simpson's method.

SECONDARY OUTCOMES:
Left ventricular end diastolic volume | week 12, and 65
  Standard transthoracic echocardiography will be performed. Left ventricular (LV) volumes will be calculated using the biplane Simpson's method.
Global longitudinal strain | week 3, 12, and 65
  Standard transthoracic echocardiography with Speckle tracking will be performed.
Left ventricular end systolic volume | week 3, 12, and 65
  Standard transthoracic echocardiography will be performed.
Left ventricular ejection fraction | week 3, 12, and 65
  Standard transthoracic echocardiography will be performed.
Pulse wave tissue Doppler imaging of the mitral annulus velocity (E') | week 3, 12, and 65
  Standard transthoracic echocardiography with tissue Doppler imaging will be performed.
Cardiac stress markers | week 3, 12, and 65
  Blood samples are analysed for markers of cardiac 'stress' (NT-pro BNP, Troponin T hs)
Peak oxygen uptake of maximal cardiopulmonary exercise test | week 1, 3, 12, and 65
  Cardiopulmonary exercise testing (CPET) will be performed on a cycle ergometer. Respiratory parameters [oxygen (O2) consumption, carbon dioxide (CO2) production] will be measured continuously.
Vascular function | week 3, 12, and 65
  Vascular function will be determined by measurement of arterial stiffness.
Leg muscle volume and function | week 3, 12, and 65
  Muscle cross-sectional area (CSA) will be assessed with peripheral computed tomography (pQCT) at the thigh.
Leg muscle function | week 3, 12, and 65
  Jumping mechanography will be performed using a mobile force plate.
Heart rate variability | week 3, 12, and 65
  Heart rate variability will be continuously recorded during 5 min in supine position and 5 min standing after an orthostatic challenge using an ECG monitor.
Quality of life | week 3, 12, and 65
  Short form quality of life questionnaire (SF36)
Quality of life with heart failure | week 3, 12, and 65
  Minnesota living with heart failure questionnaire

OTHER OUTCOMES:
Cardiac stress markers | week 4 and 12
  Blood samples for determination of markers of atrial and ventricular 'stress' (NT-pro Brain Natriuretic Peptide, Troponin T hs) are taken after a training session.
Inflammation markers | week 4 and 12
  Blood samples for determination of markers of inflammation (hs C-reactive protein, Interleukin 6) are taken after a training session.
Heart rate variability | week 4 and 12
  Heart rate variability will be continuously recorded during 5 min in supine position and 5 min standing after an orthostatic challenge in the morning following a training session.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Trachsel, MD, Principal Investigator — Preventive Cardiology & Sports Medicine, University Clinic for Cardiology, University Hospital Berne
Locations (1):
- Preventive Cardiology & Sports Medicine, University Clinic for Cardiology, University Hospital Berne, Bern, Switzerland

REFERENCES:
- [Background] Moholdt T, Aamot IL, Granoien I, Gjerde L, Myklebust G, Walderhaug L, Brattbakk L, Hole T, Graven T, Stolen TO, Amundsen BH, Molmen-Hansen HE, Stoylen A, Wisloff U, Slordahl SA. Aerobic interval training increases peak oxygen uptake more than usual care exercise training in myocardial infarction patients: a randomized controlled study. Clin Rehabil. 2012 Jan;26(1):33-44. doi: 10.1177/0269215511405229. Epub 2011 Sep 21. PMID 21937520
- [Background] Bochenek T, Wita K, Tabor Z, Grabka M, Krzych L, Wrobel W, Berger-Kucza A, Elzbieciak M, Doruchowska A, Gluza MT. Value of speckle-tracking echocardiography for prediction of left ventricular remodeling in patients with ST-elevation myocardial infarction treated by primary percutaneous intervention. J Am Soc Echocardiogr. 2011 Dec;24(12):1342-8. doi: 10.1016/j.echo.2011.09.003. Epub 2011 Oct 14. PMID 22000785
- [Background] Rognmo O, Hetland E, Helgerud J, Hoff J, Slordahl SA. High intensity aerobic interval exercise is superior to moderate intensity exercise for increasing aerobic capacity in patients with coronary artery disease. Eur J Cardiovasc Prev Rehabil. 2004 Jun;11(3):216-22. doi: 10.1097/01.hjr.0000131677.96762.0c. PMID 15179103
- [Background] Kemi OJ, Haram PM, Loennechen JP, Osnes JB, Skomedal T, Wisloff U, Ellingsen O. Moderate vs. high exercise intensity: differential effects on aerobic fitness, cardiomyocyte contractility, and endothelial function. Cardiovasc Res. 2005 Jul 1;67(1):161-72. doi: 10.1016/j.cardiores.2005.03.010. Epub 2005 Apr 20. PMID 15949480
- [Derived] Marcin T, Trachsel LD, Dysli M, Schmid JP, Eser P, Wilhelm M. Effect of self-tailored high-intensity interval training versus moderate-intensity continuous exercise on cardiorespiratory fitness after myocardial infarction: A randomised controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101490. doi: 10.1016/j.rehab.2021.101490. Epub 2021 Nov 21. PMID 33450366